CLINICAL TRIAL: NCT01504100
Title: The Effects of Distal Femoral Rotation on Patellofemoral Pain Syndrome Treated With Patella Taping
Brief Title: Efficiency of Patellar Taping in Treatment of Patellofemoral Pain Syndrome
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201103111RC
Record Dates: First submitted 2011-07-01; First posted 2012-01-05 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- femoral internal rotation
- no femoral internal rotation

SUMMARY:
Patellar subluxation is a common disorder that may cause patellofemoral pain syndrome. The efficiency of patellar taping in the treatment of patellofemoral pain syndrome has been reported good outcomes in most patients. However, some studies reported less effective in patients with higher body mass index, larger lateral patellofemoral angle, and smaller Q angle. The investigators hypothesized that femoral internal rotation is a negative factor to the patellar taping. The investigators enroll consecutive 100 patients with anterior knee pain and radiographic evidence of patellar subluxation. The investigators determine femoral rotation via physical examination. The visual analogue scale was evaluate to compare the result between the those with and without femoral internal rotation.

DETAILED DESCRIPTION:
Consecutive 100 patients with anterior knee pain and compatible with inclusion criteria. Before treatment, an independent physiotherapist evaluates whether femoral internal rotation or not via physical therapy, and another studying nurse records the visual analog scale and measures Q angle. After evaluation, McConnell taping is applied to these patients. Two weeks later, outcomes are recorded including visual analog scale, satisfactory, and complication. The outcomes are compared between those with and without femoral internal rotation.

ELIGIBILITY:
Inclusion Criteria:

* anterior knee pain
* radiographic evidence of patellar subluxation

Exclusion Criteria:

* history of patellar dislocation
* osteoarthritis of ipsilateral knee
* pregnancy
* history of knee injury
* BMI > 35
* allergy to taping

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 100 patients
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Knee pain | two weeks
  The visual analog scale are measured before and two weeks after taping.

SECONDARY OUTCOMES:
Satisfactory | 2 weeks
  The patients recorded the satisfactory score by theyself from 0 to 10. Ten degree means most satisfactory.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Chuan Jiang, MD. PhD, Study Chair — Department of Orthopaedic Surgery, National Taiwan University Hospital, 7 Chungsan South Road, Taipei, Taiwan
Locations (1):
- Department of Orthopaedic Surgery, National Taiwan University Hospital, Taipei, Taiwan